CLINICAL TRIAL: NCT07364396
Title: An Open-label, Multi-center, Single-arm Phase 1/2 Study to Assess Tolerability, Safety and Efficacy of CRC01 in Participants With Severe, Refractory Autoimmune Diseases: Systemic Lupus Erythematosus
Brief Title: Efficacy and Safety of CRC01 in Participants With Severe, Refractory Systemic Lupus Erythematosus
Acronym: CRC01-02
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Curocell Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC01-02
Record Dates: First submitted 2025-08-20; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis; Lupus Nephritis (LN); SLE; SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRC01 (Experimental): Participants with lupus nephritis will receive a single intravenous infusion of CRC01 (autologous anti-CD19 CAR-T cells) following lymphodepleting pre-conditioning chemotherapy.
  Interventions: Biological: CRC01

INTERVENTIONS:
Biological: CRC01 — Autologous T lymphocytes genetically modified to express anti-CD19 chimeric antigen receptor (CAR). Administered as a single intravenous infusion.

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of CRC01, an investigational autologous anti-CD19 chimeric antigen receptor T-cell (CAR-T) therapy, in people with lupus nephritis (LN), a serious kidney complication of systemic lupus erythematosus (SLE).

The main objectives of the study are:

1. To determine whether CRC01 infusion can improve kidney outcomes and reduce disease activity in participants with lupus nephritis.
2. To assess the safety profile, including potential risks such as cytokine release syndrome (CRS) and neurotoxicity.

Study Design This is a single-arm, open-label, multi-center, Phase 1/2 study. All enrolled participants will receive CRC01 after screening and baseline assessments.

Study Procedures

Participants will:

* Undergo eligibility screening, including blood tests, urine tests, and disease activity assessments.
* Provide autologous T lymphocytes through a procedure called leukapheresis.
* Receive a lymphodepleting pre-conditioning regimen (short course of chemotherapy).
* Receive a single intravenous infusion of CRC01 cells.
* Be hospitalized for close monitoring to detect and manage early adverse events such as CRS or neurotoxicity.
* Return for scheduled follow-up assessments through Week 52 (12 months) post-infusion to evaluate safety and treatment response.

Key Outcomes

Researchers will measure:

* Changes in proteinuria and kidney function.
* Changes in disease activity scores.
* Incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older, voluntarily provides written informed consent.
* Diagnosis of systemic lupus erythematosus (SLE) according to the 2019 EULAR/ACR classification criteria.
* Positive antinuclear antibody (ANA) at screening (titer ≥1:80).
* Diagnosis of lupus nephritis Class III or IV (with or without concurrent Class V), confirmed by kidney biopsy within 1 year prior to screening based on ISN/RPS 2018 criteria.
* Inadequate response to, or intolerance of, at least two or more standard therapies for 6 months or longer (cyclophosphamide, mycophenolate mofetil, azathioprine, tacrolimus, rituximab, belimumab).
* Proteinuria at screening with urine protein-to-creatinine ratio (UPCR) >1.5.
* Adequate laboratory values at screening: Hemoglobin >8.0 g/dL; ANC >1,000/μL; Platelets ≥50,000/μL; Total bilirubin ≤2.0 × ULN; AST and ALT ≤3 × ULN; eGFR ≥30 mL/min/1.73 m².
* Hemodynamically stable, no pericardial effusion, and LVEF ≥50% by echocardiogram at screening.
* FEV1/FVC ≥70% at screening.
* Willing and able to comply with study visits, procedures, and requirements.
* Women of childbearing potential and men must agree to use effective contraception for at least 1 year after CRC01 infusion until PCR testing confirms clearance of CRC01.

Exclusion Criteria:

* Current or anticipated requirement for renal dialysis during the study.
* History of kidney transplantation or planned transplantation during the study.
* History of severe CNS lupus or currently active severe CNS lupus.
* Prior CAR-T cell therapy.
* History of malignancy except for: basal or squamous cell carcinoma of skin treated and disease-free ≥3 years; in-situ carcinoma of cervix or breast treated and disease-free ≥3 years; superficial bladder cancer treated and disease-free ≥3 years; completely resected primary malignancy in complete remission ≥5 years.
* Unstable angina and/or myocardial infarction within 1 year prior to screening.
* Congestive heart failure of NYHA Class III or IV within 1 year prior to screening.
* Thromboembolism, pulmonary embolism, or clinically significant bleeding diathesis within 6 months prior to screening.
* Hypoxemia, clinically significant pleural effusion, or abnormal ECG findings within 6 months prior to screening.
* Stroke (ischemic or hemorrhagic) within 6 months prior to screening.
* Positive HBsAg; positive anti-HCV (eligible if HCV RNA negative); known HIV infection; or active neurological autoimmune/inflammatory diseases (e.g., Guillain-Barré syndrome, ALS).
* Recurrent or symptomatic ventricular tachycardia, or atrial fibrillation with rapid ventricular response despite therapy within 3 months prior to screening.
* Severe or uncontrolled active infection requiring systemic therapy at screening.
* Rapidly progressive disease or otherwise unsuitable for study participation, per investigator judgment.
* Pregnant or breastfeeding women.
* Known hypersensitivity to investigational product components.
* Participation in another investigational study within 4 weeks prior to screening.
* Receipt of systemic corticosteroids at therapeutic doses within 7 days prior to leukapheresis (≤7.5 mg/day prednisone equivalent is permitted).
* Receipt of immunosuppressive agents within 7 days prior to leukapheresis.
* Receipt of antibody-based therapies (e.g., belimumab, rituximab, anifrolumab) within 4 weeks prior to leukapheresis.

Inclusion Criteria for CRC01 Infusion:

* No clinically significant worsening of organ function after screening.
* If any of the following adverse events related to lymphodepleting chemotherapy exceed Grade 1 or worsen compared with screening, CRC01 infusion must be delayed:

  * Requirement for supplemental oxygen
  * New arrhythmia symptoms or clinically significant changes in cardiac function compared with screening
  * Hypotension requiring treatment
  * Active infection within 72 hours prior to the planned CRC01 infusion

    * If bacterial, viral, or fungal infection is documented, improvement of symptoms must be documented before infusion.
* Women of childbearing potential must have a negative urine pregnancy test prior to infusion.
* If CRC01 infusion is delayed for more than 2 weeks after lymphodepleting chemotherapy, administration may proceed only with approval from the sponsor's medical monitor.
* No receipt of therapeutic doses of systemic corticosteroids or immunosuppressive agents within 7 days prior to CRC01 infusion. (Prednisone ≤7.5 mg/day or equivalent is permitted.)
* No receipt of antibody-based therapies (e.g., belimumab, rituximab, anifrolumab) within 4 weeks prior to CRC01 infusion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Study: To evaluate the tolerability of CRC01 in patients with severe refractory autoimmune disease (systemic lupus erythematosus), and to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) | 28 day
  Safety and tolerability will be assessed by:
  1. Number of participants with dose-limiting toxicities (DLTs) within 28 days after CRC01 infusion, as assessed by CTCAE v5.0 and ASTCT consensus criteria.
Phase 1 Study: To evaluate the tolerability of CRC01 in patients with severe refractory autoimmune disease (systemic lupus erythematosus), and to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) | 28 day
  Safety and tolerability will be assessed by:
  2. Determination of the maximum tolerated dose (MTD) defined as the highest dose level at which ≤1 of 6 participants experience a DLT.
Phase 1 Study: To evaluate the tolerability of CRC01 in patients with severe refractory autoimmune disease (systemic lupus erythematosus), and to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) | 28 day
  Safety and tolerability will be assessed by:
  3. Determination of the recommended Phase 2 dose (RP2D) based on incidence of DLTs, safety profile, and investigator/sponsor assessment.
Phase 2 Study: To evaluate the efficacy of CRC01 by assessing Complete Renal Response (CRR) | 24 weeks
  Complete Renal Response (CRR): Defined as meeting all of the following criteria:
  1. 24-hour urine protein ≤0.5 g, or urine protein-to-creatinine ratio (UPCR) ≤0.5.
  If a 24-hour urine collection is available and meets adequacy criteria, 24-hour urine protein assessment takes precedence. If the 24-hour urine collection is inadequate or not performed, UPCR will be used for evaluation.
Phase 2 Study: To evaluate the efficacy of CRC01 by assessing Complete Renal Response (CRR) | 24 weeks
  Complete Renal Response (CRR): Defined as meeting all of the following criteria:
  2. eGFR ≥60 mL/min/1.73m², or a decrease in eGFR ≤20% compared with the pre-flare value.
Phase 2 Study: To evaluate the efficacy of CRC01 by assessing Complete Renal Response (CRR) | 24 weeks
  Complete Renal Response (CRR): Defined as meeting all of the following criteria:
  3. No use of rescue medication for systemic lupus erythematosus (SLE). (Use of corticosteroids equivalent to ≤7.5 mg/day prednisone is permitted.)

SECONDARY OUTCOMES:
Complete Renal Response (CRR) or Partial Renal Response (PRR) at each assessment Visit | Up to Week 52
  PRR is defined as ≥50% reduction in UPCR compared with baseline.
Change From Baseline in Urine Protein-to-Creatinine Ratio (UPCR) | up to Week 52
  Change from baseline in UPCR measured in urine (mg/mg)
Change From Baseline in Serum Creatinine | up to Week 52
  Change from baseline in serum creatinine. Unit of measure (mg/dL)
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) | up to Week 52
  Change from baseline in eGFR. Unit of measure: mL/min/1.73 m²
Change from baseline in UPCR, serum creatinine, urine protein, and eGFR | up to Week 52
  Composite evaluation of renal parameters including UPCR (mg/mg)
Time to achieve UPCR ≤0.5 | Up to Week 52
  Time from baseline to first achievement of UPCR ≤0.5.
Change from baseline in SLEDAI-2K scores | Weeks 12, 24, and 52
  Evaluation of change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K)
Change From Baseline in Physician's Global Assessment at Week 12 | Week 12
  Change in Physician's Global Assessment (PGA; scale 0-3)
Change From Baseline in Physician's Global Assessment at Week 24 | Week 24
  Change in Physician's Global Assessment (PGA; scale 0-3)
Change From Baseline in Physician's Global Assessment at Week 52 | Week 52
  Change in Physician's Global Assessment (PGA; scale 0-3)
Achieving LLDAS at each assessment Visit | Weeks 12, 24, and 52
  Percentage of participants achieving Low Lupus Disease Activity State (LLDAS)
Change from baseline in SF-36 scores | Weeks 12, 24, and 52
  Change in health-related quality of life assessed by Short Form Health Survey-36 (SF-36)
Change from screening in immunology parameters | up to Week 52
  Composite evaluation of immunology markers including C3, C4 (mg/dL), anti-dsDNA antibody (IU/mL), and autoantibody titers (ANA, Anti-Sm, Anti-Ro 52/60, Anti-La). Each marker will be summarized separately and reported by its corresponding unit of measure.

IPD SHARING:
Plan to Share IPD: No